CLINICAL TRIAL: NCT05101486
Title: A Randomized, Double-blind Phase 3 Study to Assess the Immunogenicity and Safety of an Ad26.RSV.PreF-based Regimen at the End of Shelf-life in Adults Aged 60 to 75 Years
Brief Title: A Study of an Ad26.RSV.PreF-based Regimen at the End of Shelf-life in Adults Aged 60 to 75 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109069; 2021-002388-23 (EudraCT Number); VAC18193RSV3003 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2021-10-29; First posted 2021-11-01 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Virus Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Ad26.RSV.PreF-based Vaccine (Experimental): Participants will receive a single intramuscular (IM) injection of Ad26.RSV.PreF-based vaccine on Day 1 (non-aged lot).
  Interventions: Biological: Ad26.RSV.PreF-based Vaccine
- Group 2: Ad26.RSV.PreF-based Vaccine (Experimental): Participants will receive a single IM injection of Ad26.RSV.PreF-based vaccine on Day 1 (aged lot 1).
  Interventions: Biological: Ad26.RSV.PreF-based Vaccine
- Group 3: Ad26.RSV.PreF-based Vaccine (Experimental): Participants will receive a single IM injection of Ad26.RSV.PreF-based vaccine on Day 1 (aged lot 2).
  Interventions: Biological: Ad26.RSV.PreF-based Vaccine

INTERVENTIONS:
Biological: Ad26.RSV.PreF-based Vaccine — Ad26.RSV.PreF-based Vaccine will be administered as single IM injection.

SUMMARY:
The purpose of this study is to demonstrate non-inferiority in terms of humoral immune responses of Ad26.RSV.preF-based study vaccine lots representative of different aged vaccine in comparison to a non-aged Ad26.RSV.preF-based study vaccine lot.

ELIGIBILITY:
Inclusion Criteria:

* Before randomization, a participant must be: a) postmenopausal (postmenopausal state is defined as no menses for 12 months without an alternative medical cause); and b) not intending to conceive by any methods
* From the time of vaccination through 3 months after vaccination, agrees not to donate blood
* In the investigator's clinical judgment, a participant must be in stable health at the time of vaccination. Participants may have underlying illnesses such as hypertension, congestive heart failure, chronic obstructive pulmonary disease, Type 2 diabetes, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms and signs are stable at the time of vaccination, and these conditions receive routine follow-up by the participant's healthcare provider. Participants will be included on the basis of medical history and vital signs performed between informed consent form (ICF) signature and vaccination
* Must be able to read, understand, and complete questionnaires in the electronic diary (eDiary)
* Must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study
* Must be able to work with smartphones/tablets/computers

Exclusion Criteria:

* Known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine)
* Abnormal function of the immune system resulting from clinical conditions or medication
* Per medical history, participant has chronic active hepatitis B or hepatitis C infection
* History of acute polyneuropathy (example, Guillain-Barré syndrome) or chronic idiopathic demyelinating polyneuropathy
* Has had major surgery (per the investigator's judgment) within 4 weeks before administration of the study vaccine or will not have recovered from surgery per the investigator's judgment at time of vaccination
* Has had major psychiatric illness and/or drug or alcohol abuse which in the investigator's opinion would compromise the participant's safety and/or compliance with the study procedures

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (13):
- United States (13):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Achieve Clinical Research, LLC, Vestavia Hills, Alabama
  - Hope Research Institute, Phoenix, Arizona
  - Clinical Research Consulting, Milford, Connecticut
  - Accel Research Sites, DeLand, Florida
  - Pharmax Research Clinic Inc, Miami, Florida
  - Suncoast Research Group, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Centennial Medical Group, Elkridge, Maryland
  - Be Well Clinical Studies, Lincoln, Nebraska
  - American Health Network, LLC, Charlotte, North Carolina
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg: Participants received adenovirus serotype 26 pre-fusion conformation-stabilized F protein (Ad26. RSV.preF) 1.0*10^11 viral particles (vp) and respiratory syncytial virus prefusion F-protein (RSV preF) 150 micrograms (mcg) mixture-based vaccine (Ad26/protein preF RSV) as intramuscular (IM) injection on Day 1.
- Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg: Participants received Ad26.RSV.preF 2.5*10^10 vp and RSV.preF protein 150 mcg mixture-based vaccine (Ad26/protein preF RSV) as IM injection on Day 1.
- Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg: Participants received Ad26.RSV.preF 1.0*10^10 vp and RSV.preF protein 150 mcg mixture-based vaccine (Ad26/protein preF RSV) as IM injection on Day 1.
Period: Overall Study
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg
Started | 251 | 252 | 252
Vaccinated (Full Analysis Set [FAS]) | 250 | 251 | 251
Completed | 231 | 241 | 228
Not Completed | 20 | 11 | 24
Not completed — Death | 1 | 0 | 1
Not completed — Lost to Follow-up | 12 | 8 | 17
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2 | 4
Not completed — Randomized but not vaccinated | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received study vaccine, regardless of the occurrence of protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg | Total
Number analyzed (Participants) | 250 | 251 | 251 | 752
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (4.37) | 65.5 (4.42) | 65.5 (4.27) | 65.6 (4.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 145 | 144 | 416
  Male | 123 | 106 | 107 | 336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 150 | 144 | 144 | 438
  Not Hispanic or Latino | 98 | 105 | 105 | 308
  Unknown or Not Reported | 2 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 39 | 42 | 41 | 122
  White | 209 | 206 | 207 | 622
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 250 | 251 | 251 | 752

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Prefusion F-protein (preF) Antibodies as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) 14 Days Post Vaccination
Description: GMTs of pre-F antibodies as assessed by ELISA at 14 days post administration of Ad26/protein preF RSV vaccine were reported.
Time Frame: 14 days post vaccination on Day 1 (Day 15)
Population: The per-protocol immunogenicity (PPI) set included all randomized participants who received the study vaccine, and for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per liter (EU/L)
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 236 | 241 | 233
ELISA units per liter (EU/L) | 4277 [3891 to 4701] | 4121 [3722 to 4562] | 4602 [4154 to 5099]

2. Secondary Outcome: Respiratory Syncytial Virus (RSV) A2 Strain Neutralizing Antibody Titers at 14 Days Post Vaccination
Description: RSV A2 strain neutralizing antibody titers of the vaccine-induced immune response was assessed through virus neutralization assay at 14 days post administration of Ad26/protein preF RSV-based vaccine were expressed as 50 percent (%) inhibitory concentration (IC50) units.
Time Frame: 14 days post vaccination on Day 1 (Day 15)
Population: The PPI set included all randomized participants who received the study vaccine, and for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 236 | 241 | 233
Titers | 6516 [5834 to 7278] | 5538 [4937 to 6212] | 6846 [6035 to 7766]

3. Secondary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) for 7 Days Post Vaccination
Description: Number of participants with solicited local AEs 7 days post vaccination were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs were precisely defined events that participants were specifically asked about and which were noted by participants in the diary. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site).
Time Frame: Up to Day 7 post vaccination on Day 1 (up to Day 8)
Population: The full analysis set (FAS) included all participants who received study vaccination, regardless of the occurrence of protocol deviations. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 243 | 248 | 247
Participants | 119 | 103 | 81

4. Secondary Outcome: Number of Participants With Solicited Systemic AEs for 7 Days Post Vaccination
Description: Number of participants with solicited systemic AEs 7 days post vaccination were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited systemic events include events such as fatigue, headache, nausea, myalgia, and pyrexia, for which participants were specifically questioned and which were noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to Day 7 post vaccination on Day 1 (up to Day 8)
Population: The FAS included all participants who received study vaccination, regardless of the occurrence of protocol deviations. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 243 | 248 | 247
Participants | 101 | 86 | 65

5. Secondary Outcome: Number of Participants With Unsolicited AEs for 28 Days Post Vaccination
Description: Number of participants with unsolicited AEs 28 days post vaccination were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant was not specifically questioned in the participant diary.
Time Frame: Up to 28 days post vaccination on Day 1 (up to Day 29)
Population: The FAS included all participants who received study vaccination, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 250 | 251 | 251
Participants | 22 | 16 | 15

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) Until 6 Months Post Vaccination
Description: Number of participants with SAEs until 6 months post vaccination were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: From Day 1 up to 6 months post vaccination on Day 1 (up to Day 183)
Population: The FAS included all participants who received study vaccination, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 250 | 251 | 251
Participants | 5 | 4 | 7

7. Secondary Outcome: Number of Participants With Adverse Event of Special Interests (AESIs) Until 6 Months Post Vaccination
Description: Number of participants with AESIs until 6 months post vaccination were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Thrombosis with thrombocytopenia syndrome (TTS) was considered as an AESI.
Time Frame: From Day 1 up to 6 months post vaccination on Day 1 (up to Day 183)
Population: The FAS included all participants who received study vaccination, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg
Number analyzed (Participants) | 250 | 251 | 251
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 until 6 months post vaccination (up to Day 183)
Description: The full analysis set (FAS) included all participants who received study vaccine, regardless of the occurrence of protocol deviations.
Arm/Group | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg
All-Cause Mortality (participants affected / at risk) | 1/250 | 0/251 | 1/251
Serious Adverse Events (participants affected / at risk) | 5/250 | 4/251 | 7/251
Other Adverse Events (participants affected / at risk) | 0/250 | 0/251 | 0/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ad26.RSV.preF 1.0*10^11 vp + RSV preF Protein 150 mcg (N=250) | Group 2: Ad26.RSV.preF 2.5*10^10 vp + RSV preF Protein 150 mcg (N=251) | Group 3: Ad26.RSV.preF 1.0*10^10 vp + RSV preF Protein 150 mcg (N=251)
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Drug Withdrawal Syndrome (General disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lung Squamous Cell Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Focal Dyscognitive Seizures (Nervous system disorders) | 0 | 1 | 0
Peroneal Nerve Palsy (Nervous system disorders) | 1 | 0 | 0
Alcohol Abuse (Psychiatric disorders) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT05101486/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT05101486/SAP_001.pdf